CLINICAL TRIAL: NCT03703141
Title: Effect of Acute or Chronic Ingestion of Sucralose on Serum Insulin in Young and Healthy Adults: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Serum Insulin Response After Acute and Chronic Sucralose Ingestion in Healthy Volunteers With Variable Body Mass Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General de México Dr. Eduardo Liceaga (Other Government)
Responsible Party: Principal Investigator, Guillermo Melendez, Projects record and follow-up chief, Hospital General de México Dr. Eduardo Liceaga
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Screening
Other Study IDs: 261575
Record Dates: First submitted 2018-07-12; First posted 2018-10-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: sucralose; insulin; AUC; young; inflammatory markers; intolerance
MeSH Terms: conditions — Insulin Resistance | interventions — trichlorosucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Sucralose 48 mg (Experimental): Sucralose 48 mg in 60 ml of water O.D. for ten weeks
  Interventions: Dietary Supplement: sucralose 48 mg (splenda)/day for ten weeks
- Sucralose 96 mg (Experimental): sucralose 96 mg in 60 ml of water O.D. for ten weeks
  Interventions: Dietary Supplement: sucralose 48 mg (splenda)/day for ten weeks
- Placebo (Placebo Comparator): 60 ml of water as placebo O.D. for ten weeks
  Interventions: Dietary Supplement: sucralose 48 mg (splenda)/day for ten weeks

INTERVENTIONS:
Dietary Supplement: sucralose 48 mg (splenda)/day for ten weeks — volunteers will take sucralose or placebo daily for 70 days
  Other Names: sucralose 96 mg (splenda)/day for ten weeks; placebo

SUMMARY:
The consumption of non-caloric sweeteners has increased worldwide; Current publications suggest its consumption associates to insulin resistance.

The present study aims to demonstrate whether acute or chronic sucralose exposure affects insulin or carbohydrate metabolism or alters systemic inflammatory markers and microbiota in young, healthy adults.

In this prospective, randomized, double-blind, placebo-controlled clinical trial, three groups will be included with 30 healthy volunteers each. Group A will receive sucralose 48 mg/ day, group B 96 mg/day and group C plain water as placebo. Subjects will be exposed to acute (one day) and chronic (seventy days) oral sucralose ingestion. After acute or chronic exposure, volunteers will undergo into an Oral Glucose Tolerance Test (OGTT), taking blood samples at -15, 0, 15, 30, 45, 60, 75, 90, 105, 120 and 180 minutes, respectively.

Areas under the curve (AUC) for insulin and glucose, will be calculated from zero to one hundred and eighty minutes as described; for C peptide, glucagon, GIP (glucose-dependent insulinotropic polypeptide) and GLP-1 (glucagon-like peptide) measure points will be at 0, 30 and 60 minutes only. Differences between one and seventy days AUC means will be compared between the three groups, adjusting for BMI. Besides, initial and final systemic inflammatory markers and inflammatory monocytes levels will be quantified and compare between acute and chronic exposure. Also, a comparison between the percentage of acute and chronic microbiome bacterial population in feces will be made.

DETAILED DESCRIPTION:
Introduction Overweight and obesity have increased along with the rate of other non-communicable diseases worldwide. At the same time, the consumption of non-caloric sweeteners (NCS) has risen considerably among the general population. Although international organizations such as Joint FAO/WHO Expert Committee on Food Additives (JECFA) has demonstrated NCS are safe; two recent publications suggested its consumption associates with insulin resistance.

Although the authors attributed the metabolic effect to changes in the composition of intestinal microbiota as a consequence of NCS ingestion, these studies lacked a robust clinical methodology, as their design were not randomized, comparative studies and the effect of NCS on systemic inflammation biomarkers were neglected.

Outcomes The present study aims to demonstrate whether acute or chronic sucralose exposure affects insulin or carbohydrate metabolism or alters systemic inflammatory markers and microbiota in young, healthy adults.

Materials and methods It is a prospective, randomized, double-blind, placebo-controlled clinical trial, comparing three groups, with 30 healthy volunteers each, who will receive daily sucralose, for seventy days. After signing off informed consent, the first group will take 48 mg sucralose diluted in 60 mL of water; the second group will receive 96 mg / 60 ml a day, while the last group will receive 60 ml of plain water as placebo.

Inclusion criteria will be either sex, age between 18 and 35 years, with a body mass index (BMI) between 18.5 and 39.0, disease free, with light or moderate physical activity before entering the study, with a HOMA ≤3.8, non-smokers, non-alcohol drinkers, agreeing not to consume neither industrial food nor beverages related to NCS during the study, having Mexican ancestry, living in the Mexico City metropolitan area and signing informed consent to participate in the study.

Exclusion criteria Any acute disease by the time of recruitment, history of Type 1 or 2 diabetes, thyroid disease, adrenal glands disease, insulinoma, malabsorption syndrome, short bowel, HIV, any cancer, liver disease, renal disease, inflammatory bowel disease, have prescribed corticosteroids in the previous three months before enrollment or undergone to bariatric surgery. Having a BMI <18.5 or >39.0, working night shifts, unable to remain at the clinic for at least 5 hours, not accepting to stop consuming industrialized food or beverages containing NCS, not accepting to stop alcohol or tobacco consumption during the study, not consenting to participate, women in childbearing potential without pregnancy control or women pregnant or breastfeeding by the time of enrollment.

Each volunteer will be instructed to drink 60 mL of fluid containing either sucralose or water, every morning before meals for seventy days. Except on day one and day 70, when they will be requested to attend the clinic after fasting at least 8 hours. Two plastic containers to carry stool sample will be provided in advance to each participant and be requested to store a stool sample. At their arrival to the clinic the stool sample will be collected and labeled. Immediately after, they will be asked to drink the corresponding dose to day one or seventy in the presence of the investigators. Once the investigational material be drinking, an Oral Glucose Tolerance Test (OGTT), will be initiated, taking blood samples at

* 15, 0, 15, 30, 45, 60, 75, 90, 105, 120 and 180 minutes, respectively. Analysis Demographics per group will be described initially. Following, areas under the curve (AUC) for insulin and glucose, will be calculated from zero to one hundred and eighty minutes, as the measure points described above; for C peptide, glucagon, GIP (glucose-dependent insulinotropic polypeptide) and GLP-1 (glucagon-like peptide) measure points will be at 0, 30 and 60 minutes only.

Mean differences of AUCs between one and seventy days will be compared between the three groups, adjusting for BMI. Besides, initial and final systemic inflammatory markers and inflammatory monocytes levels will be quantified and compared between acute and chronic exposure. Additionally, a comparison of changes between the percentage of acute and chronic microbiome population in feces will be made.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Ages between 18 and 35 years
* Must not have suffered chronic noncommunicable or infectious diseases
* Must have been practicing light-moderate physical activity before the study
* Normal insulin resistance index according to a homeostatic model value of insulin resistance (HOMA-IR) ≤ 3.8
* Must not be smokers
* They must accept not to consume industrialized foods that contain non-caloric sweeteners during their participation in the study and be agree to receive weekly telephone reminders during the protocol
* Must accept not to consume industrialized beverages containing non-caloric sweeteners during their participation in the study
* Do not consume alcoholic beverages during their participation in the study, do not have alcoholism history and have not consumed alcoholic beverages for less than two weeks before entering to the protocol
* Must have Mexican ancestry
* The volunteers, their parents and grandparents must be from Mexico city metropolitan area
* They must sign the letter of inform consent, expressing their desire to participate as volunteers in the study

Exclusion Criteria:

* People who have any kind of serious illness at the time of the selection
* People who have been diagnosed with Diabetes Mellitus type 1 or type 2
* People who have been diagnosed with thyroid disease
* People who have been diagnosed with any adrenal glands disease
* People who have been diagnosed with insulinoma
* People who have been diagnosed with malabsorption syndrome
* People with short bowel history
* People who have been diagnosed with HIV
* People who have been diagnosed with any type of neoplasia
* People who have been diagnosed with acute or chronic liver disease
* People who have been diagnosed with kidney disease with compromise on serum glucose levels
* People who have been prescribed with corticosteroid in the last 3 months before entering to the study
* People who have been prescribed with any type of antibiotic, 4 weeks prior to entering to the protocol
* People who have been prescribed with any type of non-steroidal anti-inflammatory, 4 weeks prior to entering the protocol
* People who do not accept to remain in the Clinical Pharmacology Unit during the required time to carry out the oral glucose tolerance curves (4 hours, plus the preparation time)
* People with night jobs
* People who did not accept to abstain from consuming industrialized products containing non-caloric sweeteners during their participation in the study
* People who refused to abstain from consuming industrialized beverages containing non-caloric sweeteners during their participation in the study
* People who do not accept to abstain from consuming alcoholic beverages during their participation in the study
* People who have undergone bariatric surgery before the study
* People with inflammatory bowel disease history
* People who have smoked at least 3 cigarettes per week in the last 3 months
* People who do not sign the informed consent letter to participate in the study
* Women on reproductive age without contraception therapy.
* Pregnant women
* Women who are breastfeeding at the time of evaluating their admission to the study,

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Serum insulin levels | Change the baseline serum insulin levels at 10 weeks sucralose consumption.
  To assess the effect of acute and chronic exposure to different sucralose concentrations differentiating the area under the curve levels in healthy, young volunteers, at a glucose tolerance test of 180 minutes.

SECONDARY OUTCOMES:
C-peptide serum levels. | Change the baseline serum insulin levels at 10 weeks sucralose consumption.
  To assess the effect of acute and chronic exposure to different sucralose concentrations.
Glucose-dependent insulinotropic polypeptide serum levels. | Change the baseline serum glucose-dependent insulinotropic polypeptide levels at 10 weeks sucralose consumption.
  To assess the effect of acute and chronic exposure to different sucralose concentrations.
Glucagon serum levels | Change the baseline serum glucagon levels at 10 weeks sucralose consumption.
  To assess the effect of acute and chronic exposure to different sucralose concentrations.
Glucagon-like peptide-1 serum levels | Change the baseline serum systemic inflammatory response levels at 10 weeks sucralose consumption.
  To assess the effect of acute and chronic exposure to different sucralose concentrations.
Systemic inflammatory response (pCr, Tumor Necrosis Factor , Internferon -, IL-1, IL-6, IL-12, IL-17, e IL-23 serum levels) | Change the baseline serum systemic inflammatory response levels at 10 weeks sucralose consumption.
  To assess the effect of acute and chronic exposure to different sucralose concentrations.
Inflammatory monocytes (CD14hiCD16+ CD11c+CCR2hiCX3CR1lowCD206-) serum levels. | Change the baseline serum inflammatory monocytes levels at 10 weeks sucralose consumption.
  To assess the effect of acute and chronic exposure to different sucralose concentrations.
Anti-inflammatory markers (IL-4, IL-10, e IL-13) serum levels. | Change the baseline serum anti-inflammatory markers levels at 10 weeks sucralose consumption.
  To assess the effect of acute and chronic exposure to different sucralose concentrations.
Intestinal microbiota composition. | Change the baseline intestinal microbiota composition at 10 weeks sucralose consumption.
  To assess the effect of chronic exposure to different sucralose concentrations.
Body Mass Index (BMI) | To compare the baseline body weight at 10 weeks sucralose consumption.
  To assess the effect of chronic exposure to different sucralose concentrations.
Glucose area under the curve levels | Change the baseline serum glucose levels at 10 weeks sucralose consumption.
  Influence of Body Mass Index on the glucose mean area under the curve levels with different sucralose concentrations.
C-peptide area under the curve levels | Change the baseline serum C-peptide levels at 10 weeks sucralose consumption.
  Influence of Body Mass Index on the C-peptide mean area under the curve levels with different sucralose concentrations.
Glucagon area under the curve levels | Change the baseline serum glucagon levels at 10 weeks sucralose consumption.
  Influence of Body Mass Index on the glucagon mean area under the curve levels with different sucralose concentrations.
GLP-1 area under the curve levels | Change the baseline serum GLP-1 levels at 10 weeks sucralose consumption.
  Influence of Body Mass Index on the GLP-1 mean area under the curve levels with different sucralose concentrations.
Glucose-dependent insulinotropic polypeptide area under the curve levels. | Change the baseline serum glucose-dependent insulinotropic polypeptide levels at 10 weeks sucralose consumption.
  Influence of Body Mass Index on the glucose-dependent insulinotropic polypeptide mean area under the curve levels with different sucralose concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Melendez, MD, MSc, Principal Investigator — Hospital General de Mexico Eduardo Liceaga

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Background] Garcia LM, da Silva KS, Del Duca GF, da Costa FF, Nahas MV. Sedentary behaviors, leisure-time physical inactivity, and chronic diseases in Brazilian workers: a cross sectional study. J Phys Act Health. 2014 Nov;11(8):1622-34. doi: 10.1123/jpah.2012-0423. Epub 2014 Apr 11. PMID 24732950
- [Background] Perez-Rodriguez M, Melendez G, Nieto C, Aranda M, Pfeffer F. Dietary and physical activity/inactivity factors associated with obesity in school-aged children. Adv Nutr. 2012 Jul 1;3(4):622S-628S. doi: 10.3945/an.112.001974. PMID 22798003
- [Background] Lewis HB, Forwood SE, Ahern AL, Verlaers K, Robinson E, Higgs S, Jebb SA. Personal and social norms for food portion sizes in lean and obese adults. Int J Obes (Lond). 2015 Aug;39(8):1319-24. doi: 10.1038/ijo.2015.47. Epub 2015 Apr 14. PMID 25869600
- [Background] Hernandez B, Gortmaker SL, Colditz GA, Peterson KE, Laird NM, Parra-Cabrera S. Association of obesity with physical activity, television programs and other forms of video viewing among children in Mexico city. Int J Obes Relat Metab Disord. 1999 Aug;23(8):845-54. doi: 10.1038/sj.ijo.0800962. PMID 10490786
- [Background] Stamatakis E, Hillsdon M, Mishra G, Hamer M, Marmot M. Television viewing and other screen-based entertainment in relation to multiple socioeconomic status indicators and area deprivation: the Scottish Health Survey 2003. J Epidemiol Community Health. 2009 Sep;63(9):734-40. doi: 10.1136/jech.2008.085902. Epub 2009 Apr 27. PMID 19401278
- [Background] Glazier RH, Creatore MI, Weyman JT, Fazli G, Matheson FI, Gozdyra P, Moineddin R, Kaufman-Shriqui V, Booth GL. Density, destinations or both? A comparison of measures of walkability in relation to transportation behaviors, obesity and diabetes in Toronto, Canada. PLoS One. 2014 Jan 14;9(1):e85295. doi: 10.1371/journal.pone.0085295. eCollection 2014. PMID 24454837
- [Background] National Research Council (US). The Public Health Effects of Food Deserts: Workshop Summary. Washington (DC): National Academies Press (US); 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK208019/ PMID 25032337
- [Background] Grotz VL, Munro IC. An overview of the safety of sucralose. Regul Toxicol Pharmacol. 2009 Oct;55(1):1-5. doi: 10.1016/j.yrtph.2009.05.011. Epub 2009 May 21. PMID 19464334
- [Background] Neels JG, Olefsky JM. Inflamed fat: what starts the fire? J Clin Invest. 2006 Jan;116(1):33-5. doi: 10.1172/JCI27280. PMID 16395402
- [Background] Paredes-Turrubiarte G, Gonzalez-Chavez A, Perez-Tamayo R, Salazar-Vazquez BY, Hernandez VS, Garibay-Nieto N, Fragoso JM, Escobedo G. Severity of non-alcoholic fatty liver disease is associated with high systemic levels of tumor necrosis factor alpha and low serum interleukin 10 in morbidly obese patients. Clin Exp Med. 2016 May;16(2):193-202. doi: 10.1007/s10238-015-0347-4. Epub 2015 Apr 18. PMID 25894568
- [Background] Weisberg SP, McCann D, Desai M, Rosenbaum M, Leibel RL, Ferrante AW Jr. Obesity is associated with macrophage accumulation in adipose tissue. J Clin Invest. 2003 Dec;112(12):1796-808. doi: 10.1172/JCI19246. PMID 14679176
- [Background] Papapanagiotou A, Siasos G, Kassi E, Gargalionis AN, Papavassiliou AG. Novel Inflammatory Markers in Hyperlipidemia: Clinical Implications. Curr Med Chem. 2015;22(23):2727-43. doi: 10.2174/0929867322666150520095008. PMID 25989910
- [Background] Borgeson E, Johnson AM, Lee YS, Till A, Syed GH, Ali-Shah ST, Guiry PJ, Dalli J, Colas RA, Serhan CN, Sharma K, Godson C. Lipoxin A4 Attenuates Obesity-Induced Adipose Inflammation and Associated Liver and Kidney Disease. Cell Metab. 2015 Jul 7;22(1):125-37. doi: 10.1016/j.cmet.2015.05.003. Epub 2015 Jun 4. PMID 26052006
- [Background] Walther G, Obert P, Dutheil F, Chapier R, Lesourd B, Naughton G, Courteix D, Vinet A. Metabolic syndrome individuals with and without type 2 diabetes mellitus present generalized vascular dysfunction: cross-sectional study. Arterioscler Thromb Vasc Biol. 2015 Apr;35(4):1022-9. doi: 10.1161/ATVBAHA.114.304591. Epub 2015 Feb 5. PMID 25657309
- [Result] Fakhouri TH, Kit BK, Ogden CL. Consumption of diet drinks in the United States, 2009-2010. NCHS Data Brief. 2012 Oct;(109):1-8. PMID 23102235
- [Result] Pepino MY, Tiemann CD, Patterson BW, Wice BM, Klein S. Sucralose affects glycemic and hormonal responses to an oral glucose load. Diabetes Care. 2013 Sep;36(9):2530-5. doi: 10.2337/dc12-2221. Epub 2013 Apr 30. PMID 23633524
- [Result] Suez J, Korem T, Zeevi D, Zilberman-Schapira G, Thaiss CA, Maza O, Israeli D, Zmora N, Gilad S, Weinberger A, Kuperman Y, Harmelin A, Kolodkin-Gal I, Shapiro H, Halpern Z, Segal E, Elinav E. Artificial sweeteners induce glucose intolerance by altering the gut microbiota. Nature. 2014 Oct 9;514(7521):181-6. doi: 10.1038/nature13793. Epub 2014 Sep 17. PMID 25231862
- [Result] Grotz VL, Jokinen JD. Comment on Pepino et al. Sucralose affects glycemic and hormonal responses to an oral glucose load. Diabetes care 2013;36:2530-2535. Diabetes Care. 2014 Jun;37(6):e148. doi: 10.2337/dc13-2972. No abstract available. PMID 24855176
- [Result] Hocking SL, Stewart RL, Brandon AE, Suryana E, Stuart E, Baldwin EM, Kolumam GA, Modrusan Z, Junutula JR, Gunton JE, Medynskyj M, Blaber SP, Karsten E, Herbert BR, James DE, Cooney GJ, Swarbrick MM. Subcutaneous fat transplantation alleviates diet-induced glucose intolerance and inflammation in mice. Diabetologia. 2015 Jul;58(7):1587-600. doi: 10.1007/s00125-015-3583-y. Epub 2015 Apr 22. PMID 25899451
- [Result] Fjaere E, Aune UL, Roen K, Keenan AH, Ma T, Borkowski K, Kristensen DM, Novotny GW, Mandrup-Poulsen T, Hudson BD, Milligan G, Xi Y, Newman JW, Haj FG, Liaset B, Kristiansen K, Madsen L. Indomethacin treatment prevents high fat diet-induced obesity and insulin resistance but not glucose intolerance in C57BL/6J mice. J Biol Chem. 2014 Jun 6;289(23):16032-45. doi: 10.1074/jbc.M113.525220. Epub 2014 Apr 17. PMID 24742673
- [Result] Krysiak R, Gdula-Dymek A, Okopien B. Monocyte-suppressing effect of high-dose metformin in fenofibrate-treated patients with impaired glucose tolerance. Pharmacol Rep. 2013;65(5):1311-6. doi: 10.1016/s1734-1140(13)71489-0. PMID 24399727
- [Result] Suarez-Alvarez K, Solis-Lozano L, Leon-Cabrera S, Gonzalez-Chavez A, Gomez-Hernandez G, Quinones-Alvarez MS, Serralde-Zuniga AE, Hernandez-Ruiz J, Ramirez-Velasquez J, Galindo-Gonzalez FJ, Zavala-Castillo JC, De Leon-Nava MA, Robles-Diaz G, Escobedo G. Serum IL-12 is increased in Mexican obese subjects and associated with low-grade inflammation and obesity-related parameters. Mediators Inflamm. 2013;2013:967067. doi: 10.1155/2013/967067. Epub 2013 Feb 20. PMID 23533314
- [Result] Qu HQ, Li Q, Rentfro AR, Fisher-Hoch SP, McCormick JB. The definition of insulin resistance using HOMA-IR for Americans of Mexican descent using machine learning. PLoS One. 2011;6(6):e21041. doi: 10.1371/journal.pone.0021041. Epub 2011 Jun 14. PMID 21695082
- [Result] Klein DA, Boudreau GS, Devlin MJ, Walsh BT. Artificial sweetener use among individuals with eating disorders. Int J Eat Disord. 2006 May;39(4):341-5. doi: 10.1002/eat.20260. PMID 16523474
- [Result] Allison DB, Paultre F, Maggio C, Mezzitis N, Pi-Sunyer FX. The use of areas under curves in diabetes research. Diabetes Care. 1995 Feb;18(2):245-50. doi: 10.2337/diacare.18.2.245. PMID 7729306
- [Derived] Bueno-Hernandez N, Esquivel-Velazquez M, Alcantara-Suarez R, Gomez-Arauz AY, Espinosa-Flores AJ, de Leon-Barrera KL, Mendoza-Martinez VM, Sanchez Medina GA, Leon-Hernandez M, Ruiz-Barranco A, Escobedo G, Melendez G. Chronic sucralose consumption induces elevation of serum insulin in young healthy adults: a randomized, double blind, controlled trial. Nutr J. 2020 Apr 13;19(1):32. doi: 10.1186/s12937-020-00549-5. PMID 32284053
- See also: FDA. Food Additives & Ingredients. 2015 — http://www.fda.gov/Food/IngredientsPackagingLabeling/FoodAdditivesIngredients/

DOCUMENTS (4):
  • Study Protocol (2016-01-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT03703141/Prot_000.pdf
  • Informed Consent Form: Ethics Committee Aproval (2016-03-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT03703141/ICF_001.pdf
  • Statistical Analysis Plan (2016-01-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT03703141/SAP_002.pdf
  • Informed Consent Form: Informed Consent Form signed by all the volunteers (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT03703141/ICF_003.pdf